CLINICAL TRIAL: NCT06356116
Title: Accelerated Rehabilitation Program and Functional Recovery After Direct Anterior Approach for Total Hip Arthroplasty
Brief Title: Rehabilitation After Direct Anterior Approach for Total Hip Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CMUH111-REC3-029
Record Dates: First submitted 2024-02-16; First posted 2024-04-10 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Total Hip Arthroplasty
Keywords: direct anterior approach; total hip arthroplasty; accelerated rehabilitation; telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Patients will receive the current usual care of the post-operative physical therapy following existing procedure.
  Interventions: Other: Usual care
- Accelerated rehabilitation (Experimental): Patients will have pre-operative education and quicker progress rehabilitation program, and combined with telerehabilitation until 4-week post-operation.
  Interventions: Other: Accelerated rehabilitation

INTERVENTIONS:
Other: Usual care — During hospitalization, physical therapist visits the patient once or twice on day one or two post-operative (treatments including bedside standing, ambulation, stepping, active-assisted range of motion exercises).
  Educational material will be given at discharge from hospital.
  Arms: Usual care
Other: Accelerated rehabilitation — Physical therapist visits 5 times during hospitalization, including
  1. Pre-operatively: instruction regarding range of motion exercises, use of assistive device.
  2. Post-operative day zero: bedside standing, ambulation, stepping, active-assisted range of motion exercises.
  3. Post-operative day one: visit #1 continuing the day-zero exercises;
  4. Post-operative day one: visit #2 mini-squat against wall; stair negotiation training (1/2 flight).
  5. Post-operative day two: continuing the day-zero exercises; stair negotiation (1 flight); discharge from hospital in the afternoon.
  After discharge from hospital: post-operative day three ~ week 4: telerehabilitation
  Arms: Accelerated rehabilitation

SUMMARY:
The causes for total hip arthroplasty (THA) in Taiwan include ischemic necrosis of the femoral head and degenerative osteoarthritis. Contemporary, the surgical approach for total hip replacement mostly adopts the lateral approach. However, the direct anterior approach (DAA) has gained attention gradually due to its characteristics such as muscle preservation, small surgical incision length, and few surgical complications. Nevertheless, literature lacks detailed exploration or long-term follow-up on the recovery of physical functions related to fall occurrence after this type of surgery. It limits the establishment and design of suitable post-operative rehabilitation plans. Therefore, this study aims to explore and follow-up the functional recovery in patients who undergo the DAA for hip replacement using current usual care and new-designed accelerated rehabilitation program. The proposed method involves recruiting 30 patients who will undergo the DAA for total hip replacement, who will receive the current usual care plan; and another 30 patients will receive the accelerated rehabilitation program. The assessments will be conducted before the surgery and at 2, 4, 8, and 12 weeks after the operation, evaluating hip joint function, hip abduction and flexion muscle strength, balance function, and gait performance. The statistical analysis will utilize mixed-model two-factor ANOVA, comparing the preoperative and postoperative recovery of patients undergoing the DAA with different intervention programs and at different time points. The expected outcome of this study is to enhance the understanding of the functional recovery of patients undergoing the DAA for total hip replacement in terms of hip joint function, muscle strength, balance function, and gait performance after surgery. This information will help establish the targeted DAA postoperative treatment plans, which will be practically applied to patients and compared with the current usual care to assess its effectiveness, ultimately contributing to more efficient rehabilitation plans in the future.

DETAILED DESCRIPTION:
The causes for total hip arthroplasty (THA) in Taiwan include ischemic necrosis of the femoral head and degenerative osteoarthritis. Although patients experience significant improvements in pain relief, quality of life, and physical function after the procedure, the long-term follow-up studies have found residual deficits in hip abductor muscle strength, balance function, and gait, which may result in a fear of falling or related issues. Contemporary, the surgical approach for total hip replacement mostly adopts the lateral approach. However, the direct anterior approach (DAA) has gained attention gradually due to its characteristics such as muscle preservation, small surgical incision length, and few surgical complications. Nevertheless, literature lacks detailed exploration or long-term follow-up on the recovery of physical functions related to fall occurrence, such as muscle strength and gait deviations, after this type of surgery. It limits the establishment and design of suitable post-operative rehabilitation plans. Therefore, this study aims to explore and follow-up the functional recovery in patients who undergo the DAA for hip replacement using current usual care and new-designed accelerated rehabilitation program. This study will explore the recovery in muscle strength, balance function, and gait performance of the patients before and at different postoperative time points, and also compare the differences between two groups who receive different rehabilitation programs. The proposed method involves recruiting 30 patients who will undergo the DAA for total hip replacement, who will receive the current usual care plan; and another 30 patients will receive the accelerated rehabilitation program. The assessments will be conducted before the surgery and at 2, 4, 8, and 12 weeks after the operation, evaluating hip joint function, hip abduction and flexion muscle strength, balance function, and gait performance. The statistical analysis will utilize mixed-model two-factor ANOVA, comparing the preoperative and postoperative recovery of patients undergoing the DAA with different intervention programs and at different time points. The expected outcome of this study is to enhance the understanding of the functional recovery of patients undergoing the DAA for total hip replacement in terms of hip joint function, muscle strength, balance function, and gait performance after surgery. This information will help establish the targeted DAA postoperative treatment plans, which will be practically applied to patients and compared with the current usual care to assess its effectiveness, ultimately contributing to more efficient rehabilitation plans in the future.

ELIGIBILITY:
Inclusion Criteria:

* patients who will undergo the DAA for total hip replacement due to osteoarthritis or avascular necrosis of the femoral head

Exclusion Criteria:

* no other surgery in the lower extremity in the recent year
* no auto-immune or other systemic disease that affected the ambulation ability
* can not walk independently over 10 meter due to other reason before this surgery

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional recovery questionaire | before the surgery and at 2, 4, 8, and 12 weeks after the operation
  Hip Dysfunction and Osteoarthritis Outcome Score (HOOS) to evaluate the symptoms and functional limitations. The HOOS includes 40 items with five possible responses, graded from 0 to 4 (0 points = worst possible score; 100 points = best possible score)
Maximum muscle strength | before the surgery and at 2, 4, 8, and 12 weeks after the operation
  Maximum isometric contraction of the hip abductor & flexor measured in kilogram (kg) by a hand-held dynamometer (MicroFET 2, Hoggan Scientific LLC., USA)
Quality of Life questionaire | before the surgery and at 2, 4, 8, and 12 weeks after the operation
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a self-administered questionnaire consisting of 24 items divided into 3 subscales: Pain (5 items), Stiffness (2 items), and Physical Function (17 items). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

SECONDARY OUTCOMES:
Balance function | before the surgery and at 2, 4, 8, and 12 weeks after the operation
  Biodex Balance System, Biodex Corp., USA
Gait performance | at 2, 4, 8, and 12 weeks after the operation
  Seven wireless sensors (RehaGait Basic) strapped on the waist and the lower extremities, and then walk with comfortable speed on a 10-meter walkway, forth and back. The bilateral symmetry (%) in hip flexion angle will be calculated.
Walking speed | at 2, 4, 8, and 12 weeks after the operation
  Seven wireless sensors (RehaGait Basic) strapped on the waist and the lower extremities, and then walk with comfortable speed on a 10-meter walkway, forth and back. The walking speed (m/s) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiu-Chen Lin, PhD, Principal Investigator — China Medical University, Department of Physical Therapy
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No